CLINICAL TRIAL: NCT02050373
Title: Effect of Low-level Laser Therapy on Inflammatory Mediators Release During Chemotherapy-induced Oral Mucositis: a Randomized Study
Brief Title: Low-level Laser Therapy on Inflammatory Mediators During Chemotherapy-induced Oral Mucositis
Acronym: LLLTHSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Federal University of Minas Gerais (Other); Araujo Jorge Hospital (Other)
Responsible Party: Principal Investigator, Geisa Badauy Lauria Silva, Principal investigator, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 382/2011
Record Dates: First submitted 2014-01-26; First posted 2014-01-30 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Oral Mucositis
Keywords: Mucositis; inflammation; Chemotherapy; Hematopoietic stem cell transplant; Low level laser therapy; oxidative stress
MeSH Terms: conditions — Stomatitis; Mucositis; Inflammation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-Level laser (Experimental): In the laser group, an indium phosphide, galium and aluminum (InGaAIP) diode laser (660nm, 40mW, 0.16 J, 4 J/cm2) was used to irradiate oral mucosa. Subjects received the LLLT from the first day of the conditioning regimen and continued until D+7. Laser therapy was applied by a single dentist expertise in laser irradiation. The tip touched the mucosa of the lips, right and left buccal mucosa, right and left lateral tongue, ventral tongue and buccal floor, giving a total of 10 points per region.
  Interventions: Radiation: Low-Level laser
- Control (No Intervention): In the control group, patients receive only the preventive protocol bone marrow transplant industry, consisting of mouthwashes and sodium fluoride. For ethical reasons, individuals who present oral mucositis grade 2 (WHO) will receive LLLT.

INTERVENTIONS:
Radiation: Low-Level laser — Application of laser therapy in low power mucosa jugal right and left upper and lower labial mucosa, floor of the mouth, tongue side of the right and left and belly of the tongue.
  Arms: Low-Level laser

SUMMARY:
The aim of the study is to evaluate the effect of low-level laser therapy (LLLT) on the severity of oral mucositis (OM) and inflammatory mediators (pro- and anti-inflammatory cytokines, metalloproteinases and growth factors) levels in saliva and blood; furthermore, analyze the effect of LLLT in product modulation of oxidative stress and cell damage from the oral mucosa transplant patients.

DETAILED DESCRIPTION:
This is a randomized clinical trial in which the proposed analysis will be performed from saliva samples of patients transplanted bone marrow, divided into two different groups (control and laser) and collected at different times during the hospitalization of the patient. the group laser receive prophylactic laser therapy, in order to evaluate the effects of LLLT in inflammatory mediators (cytokines pro- and anti-inflammatory) as well as their effect on modulation of oxidative stress products and cell damage (nitric oxide, myeloperoxidase, interleukin-8).

ELIGIBILITY:
Inclusion Criteria:

* Schedule to receive myeloablative conditioning regimens using chemotherapy; oral mucosa lining intact on the first day of the conditioning regimen;

Exclusion Criteria:

* Patients who presented with oral oral ulceration or erosion, active oral, viral, bacterial, or fungal infections on admission, or active oral bleeding which was uncontrollable during laser therapy or had required oral tracheal intubation during hospitalization in the HSCT Unit.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geisa BL Silva, Master, Principal Investigator — Universidade Federal de Goias; Aline C Batista, Doctor, Study Director — Universidade Federal de Goias; Daniella RN Salvador, Principal Investigator — Universidade Federal de Goias

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients admitted to the Bone Marrow Transplant Unit at Hospital Araújo Jorge/Goiás Combat Cancer Association (TMO/HAJ/ACCG), between February 2012 and July 2016.
Pre-assignment Details: The patients recruited underwent block randomization and were allocated to two groups: one which would receive the low level laser therapy protocol (LLLT group) and one which would not, only the oral hygiene guidelines described above (control group).
Groups:
- Controll: In the control group, patients receive only the preventive protocol bone marrow transplant industry, consisting of mouthwashes and sodium fluoride. For ethical reasons, individuals who present oral mucositis grade 2 (WHO) will receive LLLT.
Period: Overall Study
Arm/Group | Low-Level Laser | Controll
Started | 34 | 34
Completed | 27 | 24
Not Completed | 7 | 10
Not completed — Adverse Event | 4 | 7
Not completed — Death | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Low-Level Laser: In the laser group, an indium phosphide, galium and aluminum (InGaAIP) diode laser (660nm, 40mW, 0.16 J, 4 J/cm2) was used to irradiate oral mucosa. 27 Subjects received the LLLT from the first day of the conditioning regimen and continued until D+7. Laser therapy was applied by a single dentist expertise in laser irradiation. The tip touched the mucosa of the lips, right and left buccal mucosa, right and left lateral tongue, ventral tongue and buccal floor, giving a total of 10 points per region. Low-Level laser: Application of laser therapy in low power mucosa jugal right and left upper and lower labial mucosa, floor of the mouth, tongue side of the right and left and belly of the tongue.
- Control: In the control group, 24 patients receive only the preventive protocol bone marrow transplant industry, consisting of mouthwashes and sodium fluoride. For ethical reasons, individuals who present oral mucositis grade 2 (WHO) will receive LLLT.
- Total: Total of all reporting groups
Arm/Group | Low-Level Laser | Control | Total
Number analyzed (Participants) | 27 | 24 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (14.9) | 42 (17.8) | 41 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 15 | 11 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Severity of Oral Mucositis
Description: A trained clinical member of the team who was blind to the randomization allocation scores the degree of OM, during the hospitalization, in accordance to the World Health Organization (WHO) mucositis scale as follow: grade 0, no signs or symptoms; grade 1, painless ulcers, erythema, or mild soreness; grade 2, painful erythema, edema, or ulceration but the patient is able to eat; grade 3, mucosal damage and the patient is able to ingest only liquids; and grade 4, severe mucosa damage and the patient requires parenteral or enteral support.
Time Frame: On day of the transplant (D0), on seventh day after the transplant (D7) and discharge of the patient (HD) or until day 20 (D+20).
Population: Oral Mucositis (OM) was evaluated on admission (AD), day 7 (D+7) and hospital discharge (HD) of the all patients. The severity of OM was scored in accordance with the World Health Organization (WHO), being represented by ordinal qualitative data.
Measure: Count of Participants; unit: Participants
Groups:
- Low-Level Laser: In the laser group, an indium phosphide, galium and aluminum (InGaAIP) diode laser (660nm, 40mW, 0.16 J, 4 J/cm2) was used to irradiate oral mucosa. Subjects received the LLLT from the first day of the conditioning regimen and continued until D+7. Laser therapy was applied by a single dentist expertise in laser irradiation. The tip touched the mucosa of the lips, right and left buccal mucosa, right and left lateral tongue, ventral tongue and buccal floor, giving a total of 10 points per region. Application of laser therapy in low power mucosa jugal right and left upper and lower labial mucosa, floor of the mouth, tongue side of the right and left and belly of the tongue.
- Control: In the control group, patients receive instructions on the oral hygiene protocol (dental brushing after meals, dental flossing once a day and an alcohol-free 0.12% mouthwash twice a day). For ethical reasons, individuals who present oral mucositis grade 2 (WHO) will receive LLLT.
Arm/Group | Low-Level Laser | Control
Number analyzed (Participants) | 27 | 24
Participants
  Admission: Grade 0 | 27 | 24
  Admission: Grade 1 | 0 | 0
  Admission: Grade 2 | 0 | 0
  Admission: Grade 3 | 0 | 0
  Admission: Grade 4 | 0 | 0
  Day 7: Grade 0 | 22 | 0
  Day 7: Grade 1 | 0 | 10
  Day 7: Grade 2 | 5 | 10
  Day 7: Grade 3 | 0 | 4
  Day 7: Grade 4 | 0 | 0
  Hospital Discharge: Grade 0 | 27 | 24
  Hospital Discharge: Grade 1 | 0 | 0
  Hospital Discharge: Grade 2 | 0 | 0
  Hospital Discharge: Grade 3 | 0 | 0
  Hospital Discharge: Grade 4 | 0 | 0
Statistical Analysis 1: Comparison: Low-Level Laser vs Control; The Pearson chi-square (χ2) or Fisher's Exact tests were used, at three different times (AD, D7, HD), to analyze the oral mucositis severity in the comparison between the LLLT and control groups. Statistical analysis was not performed for each grade of oral mucositis separately; Test type: Other — For the comparison between the LLLT and control groups the Pearson chi-square (χ2) or Fisher's Exact tests were used; p < 0.05, Fisher Exact

2. Secondary Outcome: Level of Inflammatory Mediators
Description: Saliva was collected in the morning, and patients were instructed to gargle with filtered water prior to collection. All the saliva produced in a 5-min interval was collected in a sterile tube. The saliva samples were then centrifuged at 1500 rpm for 10 min, and the total volumes measured with a micropipette. The supernatant was transferred to two other sterile tubes and a phosphate-buffered saline (PBS) solution (1: 1), containing protease inhibitors (0.1 mmol/1 EDTA, 0.001 mg/ml aprotinin A, and 0.05% Tween 20) which was added to one while the other maintained its pure saliva. All aliquots were frozen at -80°C to await analysis.
Time Frame: The samples were collected at three different moments of treatment: at the time of admission (AD), on the seventh day after transplantation (D+7), and on the day of discharge (with neutrophil >0.5 × 109/l for two consecutive days) (HD).
Population: Were admitted patients had to be at least 14 years of age, scheduled for autologous or allogeneic HSCT and planned treatment consisting of a myeloablative conditioning regimen with high-dose chemotherapy (HDC), without radiotherapy. Their oral mucosal lining had to be intact, and they had to have no infectious or other associated pathologies.
Measure: Median (Inter-Quartile Range); unit: Salivary Concentration (pg/mL)
Groups:
- LLLT: Patients in the LLLT group received applications from the first day of the conditioning regimen and continued every day until the seventh post-transplant day (D+7), at approximately the same time each day. Applications were made by the same professional expert laser therapy and in compliance with all necessary biosafety protocols.
Arm/Group | LLLT | Control
Number analyzed (Participants) | 27 | 24
Salivary Concentration (pg/mL)
  CXCL-8 AD | 1733 [853 to 4057] | 185 [70 to 267]
  CXCL-8 D7 | 730 [182 to 1964] | 201 [119 to 414]
  CXCL-8 HD | 1264 [131 to 7770] | 195 [143 to 300]
  NO AD | 127 [84 to 205] | 54 [23 to 104]
  NO D7 | 68 [36 to 253] | 68 [17 to 89]
  NO HD | 80 [57 to 207] | 53 [12 to 98]
  MPO AD | 62 [59 to 62] | 60 [58 to 60]
  MPO D7 | 7 [1 to 27] | 4 [2 to 8]
  MPO HD | 61 [60 to 62] | 24 [14 to 52]
Statistical Analysis 1: Comparison: LLLT vs Control; Test type: Other — Student's t test was used to numerical variables with normal distribution. The Mann-Whitney test was used to compare the cytokine values of the two groups (control and laser). The Friedman test was used to indicate differences by comparing cytokine levels at different times of assessment within each group. The Friedman and Wilcoxon tests were used for paired analyzes of the saliva collection times in the groups. All tests were used to compare the groups at the three different times (AD, D7, HD); p < 0.05, Wilcoxon (Mann-Whitney) — p<0,05

ADVERSE EVENTS:
Time Frame: The patients was evaluated daily from the day of transplantation or infusion of bone marrow (D0) until day 20 (D+20) or discharge of the patient.
Arm/Group | Low-Level Laser | Control
All-Cause Mortality (participants affected / at risk) | 3/34 | 3/34
Serious Adverse Events (participants affected / at risk) | 4/34 | 7/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low-Level Laser (N=34) | Control (N=34)
Need for oral tracheal intubation during hospitalization (General disorders) | 3 | 7 — Need for oral tracheal intubation during hospitalization
Mental confusion (Nervous system disorders) | 1 | 0 — mental confusion

LIMITATIONS AND CAVEATS:
The clinical trials with cancer patients submitted to HSCT include difficulty in homogenizing the underlying disease and treatment protocols and the influence of the underlying disease on the blood or salivary levels of chemical mediators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No